CLINICAL TRIAL: NCT05871515
Title: 3D Ultrasound of Abdominal Aortic Aneurysm Characteristics for Predicting Aneurysm Shrinkage After Endovascular Repair
Brief Title: 3D Ultrasound of Abdominal Aortic Aneurysm Characteristics
Acronym: 3D US - EVAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1929; NL81910.091.22 (Other: CCMO)
Record Dates: First submitted 2023-04-03; First posted 2023-05-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 3D ultrasound — A 3D ultrasound is performed preoperatively to measure various aneurysm characteristics

SUMMARY:
AAA characteristics are traditionally measured with computed tomography angiography (CTA), however, three-dimensional ultrasound (3D US) is emerging as a novel imaging method for AAAs. With the use of a US contrast agent, the AAA thrombus can also be distinguished from the lumen on the 3D scans. This enables 3D visualization of the AAA and its thrombus without the need for harmful radiation and nephrotoxic contrast agents, as opposed to CTA. In in vitro measurements, 3D US has already been shown to have clinically acceptable error rate with AAA diameter and volume measurement. However, it is unclear whether this is also applicable to in vivo measurements. Therefore, the aim of this prospective study is to compare preoperative 3D US AAA characteristics as measured by 3D US with contrast enhancement (3D CEUS), 3D US without contrast enhancement (3D non-CEUS) and CTA.

ELIGIBILITY:
Inclusion Criteria:

* Unruptured infrarenal or juxtarenal abdominal aortic aneurysm (AAA);
* Scheduled for elective endovascular repair (EVAR);
* Preoperative CTA with iodine contrast available;
* Informed consent form understood and signed.

Exclusion Criteria:

* BMI>40 kg/m2
* Symptomatic AAA;
* Implanted pacemaker or ICD;
* Unable to hold breath for ≤7 seconds;
* Pregnant;
* Hypersensitivity to the active substance(s) or any of the excipients in Sonovue;
* Known right-to-left cardiac shunt;
* Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg);
* Uncontrolled systemic hypertension;
* Severe pulmonary disease (e.g. COPD GOLD 3 or 4, adult respiratory distress syndrome);
* Clinically unstable cardiac disease (recent, < 3 months, or ongoing myocardial infarction, unstable angina at rest, recent percutaneous coronary intervention, clinically worsening cardiac symptoms, severe cardiac arrhythmia's, endocarditis, etc.);
* Prosthetic valves;
* Loss of renal function (GFR < 31 mL/min), end-stage renal disease;
* End-stage liver disease;
* Sepsis;
* Hypercoagulable status, recent (< 3 months) thrombosis;
* Congestive heart failure (class III or IV);
* Psychiatric or other condition that may interfere with the study;
* Participating in another clinical study that interferes on the primary outcomes of this study;
* 3D US measurement of AAA is impossible because of bowel gasses or other causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects with an AAA who are up for EVAR treatment will be included. Participants will be recruited from the Rijnstate hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
maximum AAA diameter (mm) as measured by 3D non-CEUS, 3D CEUS and CTA | Preoperatively
  For each imaging modality, the AAA and the lumen will be segmented in specialized segmentation software. Then a centerline will be computed through the lumen and perpendicular to this line, the AAA diameters are measured. From all these diameter measurements, the maximum AAA diameter will then be computed.
AAA volume (cm^3) as measured by 3D non-CEUS, 3D CEUS and CTA | Preoperatively
  For each imaging modality, the AAA will be segmented in specialized segmentation software and then the size of the volume will be computed.
lumen volume (cm^3) as measured by 3D non-CEUS, 3D CEUS and CTA | Preoperatively
  For each imaging modality, the lumen will be segmented in specialized segmentation software and then the size of the volume will be computed.
thrombus thickness (mm) as measured by 3D non-CEUS, 3D CEUS and CTA | Preoperatively
  For each imaging modality, the thrombus will be segmented in specialized segmentation software and then the thrombus thickness will be computed.
thrombus volume (cm^3) as measured by 3D non-CEUS, 3D CEUS and CTA | Preoperatively
  For each imaging modality, the thrombus will be segmented in specialized segmentation software and then the size of the volume will be computed.

SECONDARY OUTCOMES:
Maximum AAA diameter change (mm) one-year after EVAR versus preoperative | 1 year after EVAR
  Compare the maximum AAA diameter on preoperative imaging to the maximum AAA diameter on one-year imaging (within same modality).
  Aneurysm growth is defined as a growth of 5 mm or more, aneurysm shrinkage is defined as a shrinkage of 5 mm or more and any aneurysm with a change of less then 5 mm is considered to be stable.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, prof. dr., Principal Investigator — Rijnstate hospital, Arnhem, The Netherlands
Locations (1):
- Rijnstate Hospital, Arnhem, Non US/Canada, Netherlands

IPD SHARING:
Plan to Share IPD: No